CLINICAL TRIAL: NCT03192969
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of Subcutaneous Abatacept in Combination With Glucocorticoid Treatment Compared to Glucocorticoid Monotherapy in Adults With Giant Cell Arteritis
Brief Title: A Study to Evaluate Efficacy and Safety of Subcutaneous Abatacept With Steroid Treatment Compared to Steroid Treatment Alone in Adults With Giant Cell Arteritis (GCA)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-604; 2016-002697-12 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abatacept Combination Therapy (Experimental): Abatacept subcutaneous injection (125 mg/mL prefilled syringe weekly) in combination with glucocorticoid therapy (up to 28-week taper of oral prednisone daily)
  Interventions: Drug: Abatacept; Drug: Glucocorticoid Treatment
- Placebo Monotherapy- 28 Weeks (Placebo Comparator): Glucocorticoid therapy (28-week taper of oral prednisone daily) in combination with placebo subcutaneous injection (1 mL pre-filled syringe weekly)
  Interventions: Other: Placebo; Drug: Glucocorticoid Treatment
- Placebo Monotherapy- 52 Weeks (Placebo Comparator): Glucocorticoid therapy (52 week taper of oral prednisone daily) in combination with subcutaneous placebo weekly
  Interventions: Other: Placebo; Drug: Glucocorticoid Treatment

INTERVENTIONS:
Drug: Abatacept — Abatacept subcutaneous injection, 125 mg/prefilled syringe (125 mg/mL)
  Arms: Abatacept Combination Therapy
Other: Placebo — Placebo for abatacept for subcutaneous injection in 1 mL pre-filled syringes
  Arms: Placebo Monotherapy- 28 Weeks; Placebo Monotherapy- 52 Weeks
Drug: Glucocorticoid Treatment — Glucocorticoid taper (up to 52-week or 28-week of oral prednisone/prednisolone)

SUMMARY:
To investigate the safety and efficacy of abatacept with steroid treatment in comparison to steroid treatment alone in up to a 28 week taper of steroid treatment to sustain remission of Giant Cell Arteritis in adults.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* New headache (new onset or new type of localized pain in the head)
* Elevated ESR (≥ 50 mm/h by the Westergren method) or CRP ≥ 1 mg/dL
* Temporal artery abnormality (i.e. temporal artery tenderness to palpation or decreased pulsation, unrelated to arteriosclerosis of cervical arteries)
* Temporal artery biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells
* Large vessel biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells or characteristic changes of large vessel stenosis or aneurysm secondary to GCA as seen by arteriography (Magnetic Resonance Imaging/ Magnetic Resonance Angiography), ultrasound (eg, halo sign on color duplex sonography), or CT scan
* Patients must be treated with prednisone or prednisolone of 20-60 mg/day (prednisone equivalent) and be on a dose between 20-60 mg/day for at least 2 weeks prior to enrollment into the study

Exclusion Criteria:

* Rheumatic disease other than GCA such as Takayasu's Arteritis, granulomatosis with polyangiitis (Wegener's), rheumatoid arthritis, systemic lupus erythematosus
* Patients with unilateral blindness (partial or complete) or who have unstable or recurrent visual symptoms attributable to GCA within 4 weeks of randomization
* Patients with a history of dissection of aorta
* Patients with a history of myocardial infarction, stroke or transient ischemic attack attributable to GCA within the 3 months of screening
* Patients who have been treated with intravenous ("pulse") doses of glucocorticoids defined as methylprednisolone > 1000 mg/day if given within 6 weeks of randomization
* Patients who will require oral or IV glucocorticoid treatment during the trial for conditions other than GCA
* Patients at risk of tuberculosis

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2020-06-07 (Estimated); Study Completion 2021-11-23 (Estimated)

PRIMARY OUTCOMES:
Patients in sustained remission | 40 weeks (week 12 to week 52)
  Assessment based on 2-sided stratified Cochran-Mantel-Haenszel (CMH) chi-square test, stratified by baseline glucocorticoid dose group (20-< 30, 30-< 40, 40-< 50 and 50-60 mg/day) and GCA diagnosis (New vs Relapse) at a 5% significance level. Remission is defined as the absence of clinical signs and symptoms of active disease attributable to GCA.

SECONDARY OUTCOMES:
Physician's Global Assessment of Disease Activity according to visual analog scale (VAS) | Up to 52 weeks
  measured by assessment parameters
Subject Assessment of Disease Activity according to visual analog scale (VAS) | Up to 52 weeks
  measured by assessment parameters
Short Form questionnaire-36 (SF-36) | Up to 52 weeks
  Patient reported outcome assessment
Time from Week 12 to first relapse after achieving remission | 40 weeks (week 12 to week 52)
  measured by investigator
Erythrocyte sedimentation rate (ESR) | 52 weeks
  Mean change from baseline.
C-reactive protein (CRP) | 52 weeks
  Mean change from baseline.
All adverse events and serious adverse events (AEs/SAEs) | 52 weeks
  measured by incidence of AEs and SAEs
Laboratory test abnormalities | 52 weeks
  measured by laboratory test parameters
Cmin (μg/mL): Trough level serum concentration of abatacept prior to the administration of the subcutaneous injection | 104 weeks
  measured by serum concentration
Positive abatacept response relative to baseline | 52 weeks
  A validated, sensitive, electrochemiluminescence assay (ECL) method will be used to analyze the presence of anti-abatacept antibodies in serum. Samples that are confirmed positive for antibodies specific to the CTLA4 region of abatacept will be further analyzed with a validated, in vitro, cell-based bioassay to determine whether the sera contained abatacept neutralizing activity.
Cumulative glucocorticoid dose | 52 weeks
  measured as the total glucocorticoid dose used during the treatment period
EuroQOL 5 Dimensions (EQ-5D-3L) | Up to 52 weeks
  Patient reported outcome assessment
Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue Short Form 8a | Up to 52 weeks
  Patient reported outcome assessment
Resource Utilization | Up to 52 weeks
  Assessed by the number of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (92):
- United States (13):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Fullerton, California
  - Local Institution, West Hollywood, California
  - Local Institution, Denver, Colorado
  - Local Institution, Iowa City, Iowa
  - Local Institution, Kansas City, Kansas
  - Local Institution, Rochester, Minnesota
  - Local Institution, New York, New York
  - Local Institution, Cleveland, Ohio
  - Local Institution, Dayton, Ohio
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Beaumont, Texas
- Australia (6):
  - Local Institution, Northmead, New South Wales
  - Local Institution, Auchenflower, Queensland
  - Local Institution, Woodville South, South Australia
  - Local Institution, Malvern East, Victoria
  - Local Institution, Nedlands, Western Australia
  - Local Institution, Victoria Park, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Stockerau
- Belgium (3):
  - Local Institution, Leuven
  - Local Institution, Liège
  - Local Institution, Yvoir
- Local Institution, Sofia, Sofia-Grad, Bulgaria
- Canada (3):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Trois-Rivières, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Denmark (6):
  - Local Institution, Aarhus C
  - Local Institution, Esbjerg
  - Local Institution, Glostrup Municipality
  - Local Institution, Holstebro
  - Local Institution, Odense C
  - Local Institution, Silkeborg
- Estonia (2):
  - Local Institution, Tallinn
  - Local Institution, Tartu
- France (5):
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pau
  - Local Institution, Toulouse
- Germany (10):
  - Local Institution, Berlin
  - Local Institution, Dresden
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Herne
  - Local Institution, Kirchheim
  - Local Institution, Rostock
  - Local Institution, Tübingen
  - Local Institution, W?rzburg
- Greece (3):
  - Local Institution, Athens
  - Local Institution, Larissa
  - Local Institution, Thessaloniki
- Local Institution, Dublin, Ireland
- Italy (7):
  - Local Institution, Catania
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Pavia
  - Local Institution, Prato
  - Local Institution, Torino
- Netherlands (5):
  - Local Institution, Almelo
  - Local Institution, Enschede
  - Local Institution, Groningen
  - Local Institution, Helmond
  - Local Institution, Rotterdam
- Poland (5):
  - Local Institution, Bydgoszcz
  - Local Institution, Krakow
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Romania (2):
  - Local Institution, Cluj-Napoca
  - Local Institution, Sibiu
- Local Institution, Belgrade, Serbia
- Spain (6):
  - Local Institution, Barcelona
  - Local Institution, Bilbao
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, Madrid
  - Local Institution, San Cristóbal de La Laguna
  - Local Institution, Vitoria-Gasteiz
- Sweden (3):
  - Local Institution, Stockholm
  - Local Institution, Uppsala
  - Local Institution, V?ster?s
- Switzerland (5):
  - Local Institution, Basel
  - Local Institution, Bern
  - Local Institution, Fribourg
  - Local Institution, Sankt Gallen
  - Local Institution, Z?rich
- United Kingdom (3):
  - Local Institution, Westcliff-on-Sea, Essex
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, London

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx